CLINICAL TRIAL: NCT00265057
Title: Dose Finding, Safety, Pharmacokinetic and Pharmacodynamic Study of the Vascular Targeting Agent Exherin™ (ADH-1) Administered Once Weekly in 3 Week Cycles by Intravenous Infusion in Patients With N-Cadherin Expressing, Incurable, Solid Tumors (Adherex Protocol Number AHX-01-004)
Brief Title: Study of ADH-1 Given Intravenously to Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adherex Technologies, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adherex Protocol # AHX-01-004
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Neoplasms
Keywords: Cancer;; Tumors;; Neoplasms;; Anticarcinogenic Agents;; Antineoplastic Agents;; Cadherins;; Non-Small-Cell Lung Carcinoma;; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — N-Ac-CHAVC-NH2

INTERVENTIONS:
Drug: ADH -1 (Exherin™)

SUMMARY:
N-cadherin, a protein involved in blood vessel cell binding, is increased as cancer progresses, and is on the surface of many tumor cells. ADH-1 blocks N-cadherin. This study will test the safety and effects of ADH-1 in subjects with incurable, solid tumors with a protein biomarker called N-cadherin. This study will identify the amount of ADH-1 that subjects can tolerate.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Male and female patients > or = 18 years of age with a solid tumor(s) refractory to standard curative therapy or for which no curative therapy exists. Study currently enrolling only patients with non-small cell lung cancer or advanced ovarian cancer to the safety expansion phase.
* Clinically or radiologically documented measurable disease.
* Immunohistochemical evidence of N-cadherin expression (at least 1+ positive) in archived or fresh tumor tissue
* Adequate performance status and organ function, as evidenced by hematological and biochemical blood testing and electrocardiogram (ECG)

Exclusion criteria:

* Receipt of ADH-1 prior to this clinical study
* Chemotherapy, radiotherapy, or any other investigational drug within 30 days before study entry
* History of primary brain tumors or brain metastases (known or suspected) unless any lesions have completely resolved following appropriate treatment and there has been no recurrence for at least 6 months. History of spinal cord compression. History of tumors that have shown clinically significant evidence of active bleeding (e.g., gross hemoptysis, hematemesis, hematuria, melena, or bleeding superficial tumor) within 12 weeks before study entry.
* Stroke, major surgery, or other major tissue injury within 30 days before study entry
* History of congestive heart failure, myocardial infarction, angina, life threatening arrhythmias, significant electrocardiogram (ECG) abnormalities, or known hypercoagulable states

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-06; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Instituto Europeo di Oncologia, Milan
- Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland

REFERENCES:
- See also: Adherex Technologies Inc. Corporate Homepage — http://www.adherex.com